CLINICAL TRIAL: NCT06703983
Title: Comparison of the Effect of Low Glycemic Index Diet Compared to the Classical Ketogenic Diet in Reducing the Number of Seizures in Children With Drug Resistant Epilepsy
Brief Title: Efficacy of Low Glycemic Index Diet Versus Classic Ketogenic Diet in Pediatric Epilepsy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Saman Sepehrar, Saman Sepehrar (MSc Student in Nutrition), supervised by Dr. Talebi, Pediatrician, PhD in Nutrition., Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4030150
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Seizure; Epilepsy; Drug Resistant Epilepsy
Keywords: Ketogenic diet; Classic ketogenic diet; Low glycemic index diet; LGIT; CKD; Refractory epilepsy; seizure; Drug resistant epilepsy
MeSH Terms: conditions — Seizures; Epilepsy; Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: This study is an open-label randomized clinical trial with two arms:
  Low Glycemic Index therapy (LGIT) Classic Ketogenic Diet (CKD) Each arm will include 20 participants, allocated using a block randomization process. After three months, seizure reduction outcomes will be compared between the two groups.
  All 40 participants in both arms will recieve diet for 3 months.Parents will monitor and report the impact of the dietary therapy on seizure frequency, and each participant will be categorized into one of four groups based on the reported reduction:
  1. Seizure free:No more seizures reported
  2. More than 90% seizure reduction
  3. More than 50% seizure reduction
  4. Less than 50% seizure reduction Based on previous studies, a reduction of less than 50% is considered an unsuccessful therapy.
  After three months, all 40 participants will be evaluated to determine the effectiveness of each diet in treating epilepsy and results will be analyzed and reported.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Classic Ketogenic diet (Active Comparator): This study includes two arms, with participants allocated using a blocked randomization process. In the control arm, participants will follow the Classic Ketogenic Diet (CKD), a standard dietary therapy for epilepsy.The CKD is highly restrictive, with approximately 90% of total calories derived from fat, 6% from protein, and 4% from carbohydrates and this diet is really challenging for patients to follow.
  This arm will include 20 participants with drug-resistant epilepsy for whom the ketogenic diet has been asked by a pediatric neurologist and prescribed by a registered dietitian.Participants will be followed for three months, with parents documenting seizure frequency at each monthly follow-up visit.
  At the end of the study period, seizure outcomes will be analyzed and categorized into four groups:
  Seizure-free participants. Participants with >90% seizure reduction. Participants with >50% seizure reduction. Participants with <50% seizure reduction (non-responders).
  Interventions: Other: Low Glycemic index therapy; Other: Classic Ketogenic Diet
- Low glycemic index therapy (Active Comparator): In intervention arm, patients will receive a low glycemic index diet(LGIT). The LGIT is a modified form of the ketogenic diet that restricts carbohydrate intake to sources with a glycemic index of less than 50. This diet provides approximately 60% of total calories from fat, 30% from protein, and 10% from carbohydrates.In the LGIT arm, there will be 20 participants who will follow a LGIT diet under the care of a Registered Dietitian and a Pediatric Neurologist.
  After three months, seizure outcomes will be categorized into the following groups:
  At the end of the study period, seizure outcomes will be analyzed and categorized into four groups:
  Seizure-free participants. Participants with >90% seizure reduction. Participants with >50% seizure reduction. Participants with <50% seizure reduction (non-responders). Results will be analyzed and compared with Classic Ketogenic diet which serves as the standard dietary therapy for epilepsy.
  Interventions: Other: Low Glycemic index therapy; Other: Classic Ketogenic Diet

INTERVENTIONS:
Other: Low Glycemic index therapy — In intervention arm, patients will receive a low glycemic index diet(LGIT). The LGIT is a modified form of the ketogenic diet that restricts carbohydrate intake to sources with a glycemic index of less than 50. This diet provides approximately 60% of total calories from fat, 30% from protein, and 10% from carbohydrates.In the LGIT arm, there will be 20 participants who will follow a LGIT diet under the care of a Registered Dietitian and a Pediatric Neurologist. After three months, seizure outcomes will be categorized into the following groups: At the end of the study period, seizure outcomes will be analyzed and categorized into four groups: Seizure-free participants. Participants with >90% seizure reduction. Participants with >50% seizure reduction. Participants with <50% seizure reduction (non-responders). Results will be analyzed and compared with Classic Ketogenic diet which serves as the standard dietary therapy for epilepsy.
  Other Names: LGIT
Other: Classic Ketogenic Diet — This study includes two interventions: Low Glycemic Index Therapy(LGIT) and Classic Ketogenic diet(CKD) with the CKD used as a comparison.
  There will have a total of 40 participants, randomly divided into two groups and each group would have 20 participants.
  The randomization process will use the block randomization technique and will be conducted via a website.
  Participants will first have a session with a pediatric neurologist and then meet with a Dietitian who will explain the ketogenic diet in detail for them.
  The participants in the CKD group will follow a Classic Ketogenic diet where 90% of calories come from fats, 6% from proteins, and 4% from carbohydrates.
  Patients receive the diet, and investigators will remain in online contact throughout the 3-month study, with monthly in-person visits for assessment and to ensure proper adherence to the diet.
  The primary outcome will be the reduction in seizures, as reported by the participants' parents.
  Other Names: CKD

SUMMARY:
Epilepsy is a common disease among children. Today, treating epilepsy remains a major challenge, with many children affected by this condition. According to reports, 30% of children with epilepsy do not respond well to treatment. Various methods are available for managing epilepsy, one of the most accepted therapies for this condition are dietary therapies. Numerous studies have shown that dietary therapy is an effective and can have reasonable response in treating seizure.

The most commonly used dietary intervention is the Classic Ketogenic Diet (CKD). In the CKD, approximately 90% of calories come from fat, making it a highly restrictive regimen that causes significant challenges for children to follow. Many studies have reported low adherence rates due to its difficulty, with a substantial number of patients discontinuing the diet over time.

Some studies have explored the use of the Low Glycemic Index Therapy(LGIT), another form of the ketogenic diet, in managing drug-resistant epilepsy can be successful. In the LGIT, 60% of energy is derived from fat, 30% from protein, and 10% from carbohydrates. Due to the reduced fat content and greater dietary flexibility, this diet has fewer side effects and is easier to follow. Studies have also shown higher adherence rates to LGIT compared to CKD.

Although limited research is available on LGIT, existing studies suggest that it may be as effective as CKD in treating epilepsy. Given the widespread prevalence and severe complications associated with untreated epilepsy in children, Further research into dietary therapies is crucial, as untreated epilepsy can lead to irreversible damage in children.

The aim of this study is to compare the effectiveness of the Low Glycemic Index therapy and the Classic Ketogenic Diet in epilepsy treatment. If LGIT proves to be as successful as CKD, it could be considered a suitable alternative for managing epilepsy.

In this randomized clinical trial, 40 children with drug-resistant epilepsy will be enrolled. Participants will be selected from patients referred by Pediatric Neurologists to dietitians for ketogenic diet therapy.

After obtaining informed consent, participants will be randomly assigned using a block randomization method to one of two groups: the LGIT group or the CKD group. At the end of three months, the two groups will be compared in terms of seizure frequency and duration using statistical tests. The effectiveness of LGIT relative to CKD will be reported.

DETAILED DESCRIPTION:
Epilepsy is a widespread neurological conditions in children. Recent estimates suggest that 1 in 418 children live with active epilepsy. Epilepsy can negatively impact a child's growth, learning, and development, leading to cognitive impairments, learning disabilities, developmental issues, and, in severe cases, death. Therefore, finding an effective treatment is necessary. Although many drugs have been developed for the treatment of epilepsy, one-third of patients still have drug-resistant epilepsy (DRE) that does not respond well to available epilepsy drugs.

According to the International League Against Epilepsy (ILAE), drug-resistant epilepsy(DRE) is defined as a condition in which, despite the use of at least two appropriate antiepileptic drugs at the correct dose, the epilepsy still persists and the patient continues to experience seizures.According to this definition, 30% of children with epilepsy suffer from DRE. DRE patients respond poorly to pharmacologic therapies and they need alternative therapies such as surgery, vagus nerve stimulation, and dietary therapy.

In 2018, an expert consensus committee suggested the ketogenic diet as a treatment for children with DRE based on the current scientific knowledge.In epilepsy dietary therapy, Ketogenic diet can be used. The ketogenic diet is an effective, non-invasive, and non-pharmacologic treatment for refractory childhood epilepsy. The ketogenic diet for epilepsy treatment has been used since the 1920s and in different articles. It had few to no neurotoxic effects compared to multiple anti-seizure medicines.

The ketogenic diet consists of four forms: Classic ketogenic diet, Low glycemic index therapy(LGIT), Modified Atkins diet(MAD), and MCT Ketogenic diet. According to clinical guideline of the National Institute for Health and Clinical Excellence (NICE), Ketogenic diet is a non-pharmacologic treatment for children with DRE. while the exact mechanism is still unclear, it has shown to be effective.

The classic Ketogenic diet (CKD) is usually described by the ratio of fat to carbs and protein. Mostly, a 4:1 CKD is prescribed but there are other forms like 3:1 and 2.5:1 CKD.

Although the CKD is effective in the treatment of epilepsy in many studies, most patients discontinue the diet because of its unpalatable and restrictive features specially in longer periods. To increase adherence, newer forms of the KD, such as MAD and MCTKD diet have been developed.

In LGIT, carbohydrate intake is restricted to foods with glycemic index below 50. This diet consists of 60% of calories from fat, 30% from protein, and 10 from carbohydrates.

MAD is another form of Ketogenic diet. MAD consist of 65% calories from fat, 25% of calories from protein and 10% of calories from carbohydrates (17).

In MCTKD diet, 50-70% of total energy intake is from fat, including 20-30% for MCTs and 30-40% for LCTs, with protein contributing 20-30% of calories and carbohydrates providing the remaining 20% of calories. In MCTKD most of MCT oil is derived from octanoic (C8) and decanoic (C10) fatty acids.

Various clinical trials have examined the effectiveness of various forms of ketogenic diet in treating epilepsy. Our review indicates that all studies show effectiveness of ketogenic in reducing seizures, although the degree of effectiveness varied.

This study aims to address some gaps in previous research and find out how much effective LGIT is compared to Classic Ketogenic diet.A total of 40 patients will be enrolled, with 20 participants in the CKD arm and 20 in the LGIT arm.Seizure reduction will be monitored and recorded by the parents.

At the end of the study period, seizure outcomes will be analyzed and categorized into four groups:

Seizure-free participants. Participants with >90% seizure reduction. Participants with >50% seizure reduction. Participants with <50% seizure reduction (non-responders). This study can provide valuable insights for clinicians and researchers.

ELIGIBILITY:
Inclusion Criteria:

Children between 2 and 18 years old who still have epilepsy despite receiving 2 or more medications

Children with genetic disease need to receive ketogenic diet (pyruvate dehydrogenase deficiency and GLUT-1 transporter deficiency)

Exclusion Criteria:

Parents' disapproval of the child's participation in the study Having liver and kidney diseases Doctor's disapproval based on the patient's condition Absolute contraindications to the ketogenic diet

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-27 (Actual)

PRIMARY OUTCOMES:
Seizure reduction | 3 Months
  This study consists of two arms: CKD , which has been the standard therapy for many years, and LGIT , a newer type of Ketogenic diet that has shown similar results to CKD in several published studies.
  This study aims to evaluate whether LGIT is as effective as CKD while offering a more comfortable and palatable dietary option.
  All 40 participants in both arms will recieve diet for 3 months.Parents will monitor and report the impact of the dietary therapy on seizure frequency, classifying outcomes into one of four categories:
  1. Seizure free:No seizures reported
  2. More than 90% seizure reduction
  3. More than 50% seizure reduction
  4. Less than 50% seizure reduction Based on previous studies, a reduction of less than 50% is considered an unsuccessful therapy for epilepsy treatment using dietary therapy.
  After three months, all 40 participants will be evaluated to determine the effectiveness of each diet in treating epilepsy and results will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Mashhad University of Medical Sciences, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
After study is completed, data will be analyzed and it will be available through journals and electronic databases
Supporting Information: CSR
Time Frame: starting in April 2025
Access Criteria: The results will be released in an article.